CLINICAL TRIAL: NCT01070069
Title: Prospective, Multicenter, Randomized Controlled Trial of Endovascular Aneurysm Repair Using a Bilateral Percutaneous Approach (PEVAR) vs. Standard Approach (SEVAR) Using the IntuiTrak Endovascular AAA Delivery System and the Prostar XL or Perclose ProGlide Suture-Mediated Closure System
Brief Title: Percutaneous Endovascular Aneurysm Repair (PEVAR) Trial
Acronym: PEVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-0001
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-03

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Percutaneous; Preclose; Endologix; Abbott Vascular; Endovascular; PEVAR; Stent graft; Suture mediated closure devices
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard EVAR (IntuiTrak) (Active Comparator): EVAR using standard vascular exposure for access
  Interventions: Device: SEVAR (IntuiTrak)
- PEVAR (ProGlide closure) (Experimental): Percutaneous EVAR facilitated by the ProGlide closure device
  Interventions: Device: PEVAR (ProGlide closure)
- PEVAR (ProstarXL closure) (Experimental): Percutaneous EVAR facilitated by the Prostar XL closure device
  Interventions: Device: PEVAR (Prostar XL closure)

INTERVENTIONS:
Device: PEVAR (ProGlide closure) — Percutaneous EVAR facilitated by the ProGlide closure device
  Other Names: IntuiTrak; ProGlide
  Arms: PEVAR (ProGlide closure)
Device: SEVAR (IntuiTrak) — Standard vascular exposure for access prior to EVAR
  Other Names: IntuiTrak
  Arms: Standard EVAR (IntuiTrak)
Device: PEVAR (Prostar XL closure) — Percutaneous EVAR facilitated by the Prostar XL closure device
  Other Names: IntuiTrak; Prostar XL
  Arms: PEVAR (ProstarXL closure)

SUMMARY:
To determine the safety and effectiveness of PEVAR.

DETAILED DESCRIPTION:
In >30 single center publications, percutaneous EVAR facilitated with the Prostar XL or ProGlide closure has been demonstrated to be feasible. To date, no multicenter, randomized controlled trials of the approach are available. Moreover, although the IntuiTrak System and the closure devices are commercially available in the US as FDA-approved devices, no EVAR device and no closure device is FDA approved for a totally percutaneous EVAR application.

The IntuiTrak System is indicated for the treatment of abdominal aortic aneurysms with aortic necks ranging in size from 18mm to 32mm. The System includes a 19Fr integrated introducer sheath, which is designed to reduce exchanges, and may be particularly important in a percutaneous approach. Moreover, the device is the only currently approved EVAR device with a contralateral percutaneous (9Fr) indication.

Patients with abdominal aortic aneurysm who are suitable candidates for endovascular repair using the IntuiTrak System and who meet the prospectively defined inclusion/exclusion criteria specific to the trial will be randomized to PEVAR or to standard EVAR using vascular exposure access in a ratio of 2:1. Physicians who are established experts in the field of percutaneous EVAR will participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* Informed consent form understood and signed and patient agrees to all follow-up visits
* Abdominal aortic aneurysm (AAA) with maximum diameter ≥5cm, or in the range of 4 to 5cm which has increased by 0.5cm or more in the past six months
* Have a suitable ipsilateral common femoral artery for percutaneous access using a 'Pre-close' technique as detailed in the protocol
* Anatomically eligible for the IntuiTrak System per the FDA-approved indications for use (IFU)

Exclusion Criteria:

* Life expectancy <1 year as judged by the investigator;
* Psychiatric or other condition that may interfere with the study;
* Participating in the enrollment or 30-day follow-up phase of another clinical study;
* Known allergy to any device component;
* Coagulopathy or uncontrolled bleeding disorder;
* Ruptured, leaking, or mycotic aneurysm;
* Serum creatinine (S-Cr) level >1.7 mg/dL;
* Traumatic vascular injury;
* Active systemic or localized groin infection;
* Connective tissue disease (e.g., Marfan's Syndrome);
* Renal transplant patient;
* Recent (within prior three months) cerebrovascular accident or myocardial infarction;
* Planned major intervention or surgery within 30 days following the EVAR procedure;
* Requirement for an arterial conduit at the access site;
* Morbidly obese (BMI≥40);
* Calcification throughout the common femoral artery (CFA) target area anterior wall or circumferentially or over >50% of the posterior wall;
* Femoral artery aneurysm, arteriovenous fistula or pseudoaneurysm;
* Evidence of prior common femoral artery surgery (e.g., groin incision);
* Prior clip-based vascular closure device placement in either arterial access site;
* Collagen-based vascular closure device placement in either arterial access site within the prior 90 days;
* Femoral artery needle puncture in either arterial access site within the prior 30 days;
* Hematoma at the ipsilateral arterial access site
* Significant scarring at the ipsilateral arterial access site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2010-04-13 (Actual); Primary Completion 2012-03-09 (Actual); Study Completion 2012-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, MD, Principal Investigator — Endologix
Locations (20):
- United States (20):
  - Loma Linda VA Medical Center, Loma Linda, California
  - VA San Diego, San Diego, California
  - Holy Cross Medical Center, Fort Lauderdale, Florida
  - VA Gainesville, Gainesville, Florida
  - VA Miami, Miami, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Mercy Hospital, Chicago, Illinois
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Mission Hospital, Asheville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Lake Health, Willoughby, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - North Central Heart Hospital, Sioux Falls, South Dakota
  - Dallas VA Medical Center, Dallas, Texas
  - St. Luke's Hospital at Texas Heart Institute, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax, Falls Church, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Wang Q, Wu J, Ma Y, Zhu Y, Song X, Xie S, Liang F, Gimzewska M, Li M, Yao L. Totally percutaneous versus surgical cut-down femoral artery access for elective bifurcated abdominal endovascular aneurysm repair. Cochrane Database Syst Rev. 2023 Jan 11;1(1):CD010185. doi: 10.1002/14651858.CD010185.pub4. PMID 36629152
- [Derived] Nelson PR, Kracjer Z, Kansal N, Rao V, Bianchi C, Hashemi H, Jones P, Bacharach JM. A multicenter, randomized, controlled trial of totally percutaneous access versus open femoral exposure for endovascular aortic aneurysm repair (the PEVAR trial). J Vasc Surg. 2014 May;59(5):1181-93. doi: 10.1016/j.jvs.2013.10.101. Epub 2014 Jan 17. PMID 24440678
- [Derived] Krajcer Z, Nelson P, Bianchi C, Rao V, Morasch M, Bacharach J. Percutaneous endovascular abdominal aortic aneurysm repair: methods and initial outcomes from the first prospective, multicenter trial. J Cardiovasc Surg (Torino). 2011 Oct;52(5):651-9. Epub 2011 Jul 28. PMID 21796092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 Roll-in patients were entered in the study. 151 patients were randomized to either PEVAR ProGlide, PEVAR Prostar XL or SEVAR treatment for AAA repair. The enrollment period was from July 15, 2010 to February 9, 2012. The final patient completed the study in September 2012.
Pre-assignment Details: 151 Randomized patients and 41 Roll-in patients were enrolled in the study.
Groups:
- PEVAR (Prostar XL Roll-In Phase): Percutaneous EVAR facilitated by the Prostar XL closure device
  PEVAR (Prostar XL closure): Percutaneous EVAR facilitated by the Prostar XL closure device
- PEVAR (ProGlide Roll-In Phase): Percutaneous EVAR facilitated by the ProGlide closure device
  PEVAR (ProGlide closure): Percutaneous EVAR facilitated by the ProGlide closure device
Period: Overall Study
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (Prostar XL Roll-In Phase) | PEVAR (ProGlide Roll-In Phase)
Started | 50 | 50 | 51 | 19 | 22
Completed | 44 | 48 | 45 | 19 | 18
Not Completed | 6 | 2 | 6 | 0 | 4
Not completed — Death | 1 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 4 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- SEVAR: Standard vascular exposure cutdown approach (SEVAR=Control).
- PEVAR Perclose ProGlide: PEVAR performed with the Perclose ProGlide suture mediated closure system.
- PEVAR Prostar XL; PEVAR (Prostar XL Roll -In); PEVAR (ProGlide Roll -In): PEVAR performed with the Prostar XL suture mediated closure system.
- Total: Total of all reporting groups
Arm/Group | SEVAR | PEVAR Perclose ProGlide | PEVAR Prostar XL | PEVAR (Prostar XL Roll -In) | PEVAR (ProGlide Roll -In) | Total
Number analyzed (Participants) | 50 | 50 | 51 | 19 | 22 | 192
Age, Continuous [Median (Standard Deviation); unit: years] | 73 (8.8) | 70 (6.6) | 74 (10.6) | 73 (7.0) | 71 (6.9) | 72.2 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 7 | 1 | 1 | 17
  Male | 45 | 47 | 44 | 18 | 21 | 175
Race/Ethnicity, Customized [Number; unit: participants]
  White | 47 | 46 | 44 | 15 | 20 | 172
  Non-white | 3 | 4 | 7 | 4 | 2 | 20
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 51 | 19 | 22 | 151
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 28 (4.7) | 29 (3.9) | 28 (4.7) | 27 (4.4) | 29 (5.8) | 28.2 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success as Defined as the Composite of Procedural Technical Success, Absence of Vascular Complications, and Absence of Major Adverse Events as Determined by the Independent Clinical Events Committee (CEC).
Description: The primary endpoint for the trial is 30-day Treatment Success, defined as the composite of the following as determined by the independent physician adjudicator:
  * Procedural technical success
  * Absence of vascular complication
  * Absence of major adverse event
Time Frame: 30 days
Population: PEVAR (Prostar XL Roll-in) and PEVAR (ProGlide Roll-in) were not part of the primary endpoint analysis cohort and hence not included in this section.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure)
Number analyzed (Participants) | 50 | 50 | 51
Participants
  Subjects with Treatment Success | 39 | 44 | 40
  Subjects with unsuccessful Treatment | 11 | 6 | 11

2. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: SAEs for Standard EVAR, PEVAR (ProGlide closure), PEVAR (ProstarXL closure), PEVAR (ProGlide Roll-in) ,PEVAR (ProstarXL Roll-in).
Time Frame: 30 days
Population: SAEs Standard EVAR, PEVAR (ProGlide closure), PEVAR (ProstarXL closure), PEVAR (ProGlide Roll-in) ,PEVAR (ProstarXL Roll-in).
Measure: Number; unit: participants
Groups:
- PEVAR (ProGlide Roll-in): PEVAR performed with the ProGlide suture mediated closure system.
- PEVAR (ProStar XL Roll-in): PEVAR performed with the ProStar XL suture mediated closure system.
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll-in) | PEVAR (ProStar XL Roll-in)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
participants
  Patients with at least 1 SAE | 13 | 5 | 16 | 6 | 9
  Blood and lymphatic system disorders | 3 | 1 | 1 | 1 | 2
  Gastrointestinal disorders | 1 | 0 | 1 | 1 | 0
  General disorders and administration site conditions | 1 | 1 | 3 | 2 | 2
  Investigations | 4 | 3 | 2 | 0 | 0
  Nervous system disorders | 3 | 0 | 1 | 0 | 0
  Renal and urinary disorders | 2 | 2 | 4 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 2 | 0 | 2 | 1 | 1
  Vascular disorders | 4 | 0 | 4 | 2 | 4
  Infections and infestations | 0 | 1 | 3 | 0 | 0
  Metabolism and nutrition disorders | 0 | 1 | 1 | 1 | 1
  Cardiac disorders | 0 | 0 | 2 | 1 | 0
  Injury, poisoning and procedural complications | 0 | 0 | 1 | 0 | 3
  Surgical and medical procedures | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: SF-36 (Health-related Quality of Life Survey)
Description: Health-related Quality of Life per the standardized short form 36-item survey [SF-36]); self-reported groin pain per a Pain Scale.
  It comprises 36 questions which cover eight domains of health:
  1. Physical Function (Range 0 to 100)
  2. Social Functioning (Range 0 to 100)
  3. Role Limitations due to physical Health (Range o to 100)
  4. Pain (Range 0 to 100)
  5. Mental Health (Range 0 to 100)
  6. Role limitations due to emotional health (Range 0 to 100)
  7. Energy and fatigue (Range 0 to 100)
  8. General health (Range 0 to 100)
  Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 30 days
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll-in) | PEVAR (Prostar XL Roll-in)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
Scores on a Scale
  Physical Function at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  Physical Function at 1 Month | 64 (27) | 71 (27) | 60 (26) | 58 (26) | 70 (21)
  Role Limitations due to Physical Health at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  Role Limitations due to Physical Health at 1 Month | 47 (46) | 59 (40) | 51 (45) | 51 (44) | 43 (41)
  Role Limitations due to Emotional Health at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  Role Limitations due to Emotional Health at 1 Month | 72 (42) | 68 (40) | 78 (38) | 67 (44) | 79 (34)
  Energy/Fatigue at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  Energy/Fatigue at 1 Month | 54 (24) | 55 (25) | 51 (21) | 52 (25) | 63 (20)
  Mental Health at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  Mental Health at 1 Month | 79 (19) | 73 (20) | 82 (15) | 82 (17) | 87 (19)
  Social Functioning at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  Social Functioning at 1 Month | 52 (16) | 55 (17) | 53 (20) | 78 (26) | 84 (25)
  Pain at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  Pain at 1 Month | 74 (23) | 69 (27) | 78 (26) | 73 (26) | 80 (29)
  General Health at 1 Month: number analyzed (Participants) | 49 | 50 | 49 | 22 | 19
  General Health at 1 Month | 46 (16) | 48 (14) | 48 (18) | 65 (24) | 77 (15)

4. Secondary Outcome: Clinical Utility Measures
Description: In-hospital evaluations: Time in ICU; Time to ambulation; Time to normal diet; Times to possible and actual hospital discharge.
Time Frame: From Procedure to Discharge Visit
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll-in) | PEVAR (Prostar XL Roll-in)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
Hours
  ICU Length of Stay, hours: number analyzed (Participants) | 24 | 35 | 14 | 22 | 19
  ICU Length of Stay, hours | 35 (38) | 26 (9.0) | 31 (15) | 33 (11) | 12 (25)
  Time to Ambulation, hours: number analyzed (Participants) | 50 | 50 | 48 | 22 | 19
  Time to Ambulation, hours | 19 (16) | 17 (7.2) | 16 (9.1) | 22 (13) | 19 (14)
  Time to Normal Diet, hours: number analyzed (Participants) | 50 | 49 | 50 | 22 | 19
  Time to Normal Diet, hours | 15 (22) | 14 (9.4) | 10 (8.4) | 17 (7.4) | 18 (11)

5. Secondary Outcome: Clinical Utility Measures
Description: % requiring Foley catheter, central venous catheter, or gastric tube; % discharged to skilled nursing facility (SNFs) or assistive living facility (ALFs); % requiring analgesic for groin pain.
Time Frame: From Procedure to Discharge Visit
Population: All available data has been reported.
Measure: Number; unit: percentage of participants
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll-in) | PEVAR (Prostar XL Roll-in)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
percentage of participants
  Foley Catheter: number analyzed (Participants) | 41 | 40 | 38 | 21 | 17
  Foley Catheter | 82 | 80 | 80 | 96 | 89
  Central Venous Catheter: number analyzed (Participants) | 10 | 19 | 7 | 4 | 2
  Central Venous Catheter | 20 | 38 | 38 | 18 | 11
  Nasogastric Tube: number analyzed (Participants) | 3 | 7 | 1 | 3 | 19
  Nasogastric Tube | 6.0 | 14 | 2.0 | 14 | 0
  Discharged to SNF/ALF: number analyzed (Participants) | 1 | 50 | 51 | 1 | 19
  Discharged to SNF/ALF | 2.0 | 0 | 0 | 4.5 | 0

6. Secondary Outcome: Number of Participants With All Non-serious Adverse Events
Description: Adverse Events: Number of Participants with All non-serious adverse events in the three arms listed below.
Time Frame: 30 Days
Measure: Number; unit: Number of participants
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll-in) | PEVAR (Prostar XL Roll-in)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
Number of participants
  Blood and lymphatic system disorders | 3 | 1 | 3 | 4 | 2
  Gastrointestinal disorders | 6 | 9 | 4 | 2 | 5
  General disorders and administration site conditions | 19 | 12 | 10 | 13 | 9
  Infections and infestations | 4 | 4 | 2 | 1 | 0
  Injury, poisoning and procedural complications | 10 | 13 | 10 | 4 | 5
  Investigations | 16 | 23 | 19 | 11 | 5
  Metabolism and nutrition disorders | 3 | 14 | 2 | 3 | 2
  Musculoskeletal and connective tissue disorders | 2 | 0 | 3 | 1 | 2
  Nervous system disorders | 2 | 4 | 2 | 1 | 1
  Psychiatric disorders | 2 | 1 | 0 | 1 | 0
  Renal and urinary disorders | 3 | 3 | 0 | 0 | 4
  Respiratory, thoracic and mediastinal disorders | 2 | 3 | 2 | 0 | 1
  Skin and subcutaneous tissue disorders | 2 | 2 | 0 | 1 | 0
  Surgical and medical procedures | 2 | 2 | 3 | 0 | 0
  Vascular disorders | 7 | 4 | 1 | 1 | 1
  Cardiac disorders | 0 | 1 | 2 | 1 | 0
  Congenital, familial and genetic disorders | 0 | 0 | 1 | 0 | 0
  Reproductive system and breast disorders | 0 | 0 | 1 | 0 | 1

7. Secondary Outcome: Clinical Utility Measure
Description: In-hospital evaluations: Contrast media volume used
Time Frame: Through Pre-Discharge Visit
Measure: Mean (Standard Deviation); unit: mL
Groups:
- PEVAR (ProGlide Roll -In): PEVAR performed with the ProGlide suture mediated closure system.
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll -In) | PEVAR (Prostar XL Roll -In)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
mL | 144 (90) | 120 (78) | 123 (56) | 157 (94) | 118 (54)

8. Secondary Outcome: Clinical Utility Measures
Description: In-hospital evaluations: Anesthesia time; Fluoroscopy time; Time to hemostasis.
Time Frame: During Procedure
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: Min
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll -In) | PEVAR (Prostar XL Roll -In)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
Min
  Anesthesia Time, min | 203 (93) | 181 (65) | 152 (56) | 201 (75) | 2.9 (1.28)
  Fluoroscopy Time, min | 24 (14) | 26 (16) | 22 (8.5) | 30 (16) | 25 (13)
  Ipsilateral Time to Hemostasis, min | 23 (23) | 9.8 (17) | 13 (19) | 7.7 (6.8) | 5.6 (6.1)

9. Secondary Outcome: Clinical Utility Measures
Description: In-hospital evaluations: Times to possible and actual hospital discharge.
Time Frame: Through Pre-Discharge Visit
Population: All available data has been reported.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (ProGlide Roll-in) | PEVAR (Prostar XL Roll-in)
Number analyzed (Participants) | 50 | 50 | 51 | 22 | 19
Days
  EligibleTime to Hospital Discharge, days | 1.76 (2.47) | 1.2 (0.7) | 1.29 (0.83) | 1.3 (0.5) | 1.4 (1.0)
  Actual Time to Hospital Discharge, days | 1.8 (2.4) | 1.3 (0.7) | 1.4 (0.9) | 1.4 (0.5) | 2.1 (0.0)

ADVERSE EVENTS:
Time Frame: 1 Year
Description: All Adverse Events were monitored/assessed without regard to the specific adverse event term.
Arm/Group | Standard EVAR (IntuiTrak) | PEVAR (ProGlide Closure) | PEVAR (ProstarXL Closure) | PEVAR (Prostar XL Roll -In) | PEVAR (ProGlide Roll -In)
Serious Adverse Events (participants affected / at risk) | 20/50 | 13/50 | 19/51 | 9/19 | 6/22
Other Adverse Events (participants affected / at risk) | 42/50 | 44/50 | 39/51 | 14/19 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard EVAR (IntuiTrak) (N=50) | PEVAR (ProGlide Closure) (N=50) | PEVAR (ProstarXL Closure) (N=51) | PEVAR (Prostar XL Roll -In) (N=19) | PEVAR (ProGlide Roll -In) (N=22)
Blood and Lymph Disorder (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Cardiac Disorder (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
GI Disorder (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (4) | 0 (0) | 1 (1)
General Disorder (General disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Infections and Infestations (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Injury and Procedural Complications (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 6 (6) | 3 (3) | 0 (0)
Investigations (Investigations) | 4 (6) | 3 (5) | 2 (3) | 0 (0) | 0 (0)
Metabolism/Nutrition Disorders (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and Urinary Disorders (Renal and urinary disorders) | 2 (2) | 2 (3) | 6 (6) | 0 (0) | 0 (0)
Respiratory/Thoracic Disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Vascular Disorders (Vascular disorders) | 6 (7) | 1 (2) | 6 (7) | 4 (4) | 2 (2)
Surgical/Medical procedure (Surgical and medical procedures) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard EVAR (IntuiTrak) (N=50) | PEVAR (ProGlide Closure) (N=50) | PEVAR (ProstarXL Closure) (N=51) | PEVAR (Prostar XL Roll -In) (N=19) | PEVAR (ProGlide Roll -In) (N=22)
Blood and Lymph Disorders (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 4 (4) | 2 (3) | 4 (4)
Cardiac Disorders (Cardiac disorders) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Eye Disorders (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GI Disorders (Gastrointestinal disorders) | 7 (10) | 10 (12) | 4 (5) | 5 (7) | 2 (2)
General Disorders (General disorders) | 20 (27) | 12 (15) | 12 (19) | 9 (15) | 13 (16)
Infections and Infestations (Infections and infestations) | 4 (4) | 6 (8) | 3 (4) | 0 (0) | 1 (1)
injury and Procedural Complications (Injury, poisoning and procedural complications) | 17 (17) | 19 (21) | 18 (21) | 5 (6) | 4 (5)
Investigations (Investigations) | 23 (36) | 31 (54) | 24 (43) | 5 (10) | 11 (23)
Metabolism/Nutritional Disorders (Metabolism and nutrition disorders) | 4 (4) | 14 (16) | 3 (5) | 2 (5) | 3 (3)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 3 (3) | 5 (5) | 3 (3) | 1 (2) | 1 (1)
Psychiatric Disorders (Psychiatric disorders) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Renal and Urinary Disorders (Renal and urinary disorders) | 4 (4) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Reproductive Disorders (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Respiratory/Thoracic Disorders (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (8) | 2 (2) | 1 (3) | 0 (0)
Skin Disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Surgical/Medical Procedures (Surgical and medical procedures) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Vascular Disorders (Vascular disorders) | 8 (8) | 5 (6) | 8 (9) | 1 (1) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 4 (7) | 2 (2) | 1 (1)
Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other